CLINICAL TRIAL: NCT03507842
Title: A Prospective Randomized Comparison of High-dose Cytarabine an High-dose Daunorubicin in the Induction Chemothrapy for Acute Myeloid Leukemia
Brief Title: A Prospective Randomized Comparison of HDAC Vs AD in the Induction Chemothrapy for AML.
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Je-Hwan Lee, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_HDAC vs AD in AML
Record Dates: First submitted 2018-04-04; First posted 2018-04-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: HDAC vs AD
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose cytarabine (Experimental): High-dose cytarabine 3.0 g/m2 q12hr 3-hour iv infusion on days 1, 3, 5 plus daunorubicin 45 mg/m2/day continuous iv infusion for 3 days (D1-3).
  Interventions: Drug: High dose Cytarabine
- high-dose daunorubicin (Experimental): cytarabine 200 mg/m2/day continuous iv infusion for 7 days (D1-7) plus high-dose daunorubicin 90 mg/m2/day continuous iv infusion for 3 days (D1-3).
  Interventions: Drug: Cytarabine; Drug: Hign dose Daunorubicin

INTERVENTIONS:
Drug: High dose Cytarabine — High dose Cytarabine 3.0 g/m2 q12hr 3-hour iv infusion on days 1, 3, 5 plus daunorubicin 45 mg/m2/day continuous iv infusion for 3 days (D1-3).
  Other Names: HDAC
  Arms: High-dose cytarabine
Drug: Cytarabine — cytarabine 200 mg/m2/day continuous iv infusion for 7 days (D1-7)
  Other Names: AD
  Arms: high-dose daunorubicin
Drug: Hign dose Daunorubicin — Hign dose Daunorubicin 90 mg/m2/day continuous iv infusion for 3 days (D1-3).
  Other Names: AD
  Arms: high-dose daunorubicin

SUMMARY:
This trial is a single-center, non-blind, two-arm randomized prospective controlled trial to compare the effectiveness of two induction chemotherapy regimens (high-dose cytarabine plus daunorubicin [HDAC] vs. cytarabine plus high-dose daunorubicin [AD]) in acute myeloid leukemia (AML). The primary hypothesis of the study is that AD is superior to HDAC in terms of event-free survival (EFS, time from registration to induction failure, relapse, or death).

DETAILED DESCRIPTION:
* Induction chemotherapy

  * Arm I [HDAC]: cytarabine 3.0 g/m2 q12hr 3-hour iv infusion on days 1, 3, 5 plus daunorubicin 45 mg/m2/day continuous iv infusion for 3 days (D1-3).
  * Arm II [AD]: cytarabine 200 mg/m2/day continuous iv infusion for 7 days (D1-7) plus daunorubicin 90 mg/m2/day continuous iv infusion for 3 days (D1-3).
* Interim bone marrow examination Interim bone marrow aspiration and biopsy will be done between 14 and 21 days after start of induction chemotherapy. If bone marrow has blasts < 10%, no additional chemotherapy will be given until the recovery of blood counts (absolute neutrophil counts rise over 1,000/μL and platelet counts over 100,000/μL) or post-induction day 35, when bone marrow examination will be repeated to evaluate CR. After the marrow examination, re-induction course will be given. If interim bone marrow examination shows persistent leukemia (blasts ≥ 10%), re-induction course could be given. Patients who did not attain CR after the re-induction chemotherapy will be eliminated from the study.
* Re-induction chemotherapy

  * Cytarabine 200 mg/m2/day iv infusion for 5 days (D1-5) plus daunorubicin 45 mg/m2/day iv infusion for 2 days (D1-2) Post-remission consolidation chemotherapy
  * Adverse risk group: up to 3 courses of intermediate-dose cytarabine (1.0 g/m2/day iv for 5 days [D1-5]) plus etoposide (150 mg/m2/day iv for 3 days [D1-3])
  * Favorable/intermediate risk group: up to 3 courses of high-dose cytarabine (3.0 g/m2/day q12 hr iv for 3 days [D1, 3, 5])
  * Autologous or allogeneic hematopoietic cell transplantation (HCT) can be performed based on the risk of relapse.
  * The bone marrow examination will be done after the completion of consolidation chemotherapy or before HCT.

ELIGIBILITY:
Inclusion Criteria:

* Previously-untreated AML (≥ 20% blasts in bone marrow and/or peripheral blood)
* Age of 15 years or older, 60 years or younger
* Adequate performance status (Karnofsky score of 50 or more)
* Adequate hepatic and renal function (AST, ALT, and bilirubin < 2.5 x upper normal limit and creatinine < 2.0 mg/dL & creatinine clearance ≥ 50 mL/min). Elevation of AST or ALT due to hepatic infiltration of leukemic cells will be permitted.
* Adequate cardiac function (left ventricular ejection fraction ≥45% on heart scan or echocardiogram)
* Signed informed consent

Exclusion Criteria:

* Patients with history of chemotherapy for leukemia or cytarabine and anthracycline treatment for any malignancy. Hydroxyurea for reduction of leukemic cell burden before induction chemotherapy will be permitted.
* Patients with acute promyelocytic leukemia
* Patients with blast crisis of chronic myeloid leukemia
* Patients with central nervous system (CNS) leukemia or granulocytic sarcoma without bone marrow involvement
* Presence of uncontrolled and/or severe medical condition (infection, bleeding, cardiovascular disease including myocardial infarction within previous 6 months.)
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse | 3 years
  defined for all patients achieving CR; measured from the date of CR achievement until the date of relapse; patients not known to have relapsed are censored on the date they were last examined; patients who died without relapse are counted as a competing cause of failure

SECONDARY OUTCOMES:
Event-free survival | 3years
  Defined for all patients; measured from the starting date of registration to the date of induction treatment failure, or relapse from CR, or death from any cause; patients not known to have any of these events are censored on the date they were examined
Overall survival | 3years
  Defined for all patients; measured from the starting date of registration to the date of death from any cause-patients not known to have died at last follow-up are censored on the date they were last known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Je-Hwan Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No